CLINICAL TRIAL: NCT07283640
Title: A Phase IB Trial of Subcutaneous Blinatumomab in Combination With Revumenib for Patients With KMT2A-rearranged Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry); Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0932; NCI-2025-09116 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Blinatumomab; Revumenib; Lymphoblastic Leukemia; KMT2A-rearranged
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — revumenib; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Treatment with SC Blinatumomab + Revumenib in R/R ALL
  Interventions: Drug: Revumenib; Drug: Blinatumomab
- Cohort 2 (Experimental): Treatment with SC Blinatumomab + Revumenib in Newly Diagnosed ALL
  Interventions: Drug: Revumenib; Drug: Blinatumomab

INTERVENTIONS:
Drug: Revumenib — Given by po
Drug: Blinatumomab — Given by IV

SUMMARY:
To learn about the safety and effects of revumenib in combination with blinatumomab in patients with newly diagnosed or relapsed/refractory Ph-negative ALL with a KMT2A rearrangement.

DETAILED DESCRIPTION:
Primary Objectives

* To determine the safety of recommended dose by 20 participants including 10 relapsed/refractory participants (cohort 1) and 10 newly diagnosed participants (cohort 2).
* To evaluate the overall response rate (combination of complete remission [CR] + complete remission with incomplete count recovery [CRi) + complete remission with incomplete hematologic recovery [CRh]) of the combination of SC blinatumomab and revumenib in cohort 1 and cohort 2 (participants with MRD-only disease will not be included towards the overall response rate)
* To evaluate event-free survival (EFS, defined as the time from treatment initiation to relapse, death, or documented treatment failure) in cohort 2

Secondary Objectives

* To evaluate overall survival (OS, defined as the time from treatment initiation to death from any cause)
* To summarize the safety of the combination of revumenib and SC blinatumomab at all revumenib doses tested
* To evaluate measurable residual disease (MRD) negativity by flow cytometry (sensitivity of 10-4) and ClonoSeq NGS (sensitivity of 10-6)
* To characterize the frequency of lineage switch after treatment with the combination of revumenib and SC blinatumomab

ELIGIBILITY:
Eligibility Criteria

• The following groups of participants will be eligible:

* Participants > 18 years of age with relapsed and/or refractory (defined as >5% blasts in the peripheral blood or bone marrow) KMT2A-r B-cell ALL or
* Participants >18 years of age with persistent measurable residual disease by flow cytometry or next generation sequencing KMT2A-r B-cell ALL or
* Newly diagnosed participants with KMT2A-r B-cell ALL > 60 years old or unfit for intensive chemotherapy

Unfit for intensive chemotherapy defined as:

* ECOG >2
* Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction <50%, or chronic stable angina)
* Severe pulmonary disorder (e.g., DLCO <65% or FEV1 <65%)
* Creatinine clearance <45 ml/min
* Hepatic disorder with total bilirubin 1.5 x upper limit of normal
* Performance status <2 per ECOG scale (for R/R participants)
* Adequate liver function as defined by the following criteria:

  * Total serum bilirubin <1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 x ULN
* Adequate pancreatic function as define by serum lipase and amylase < 1.5 x ULN
* For females of childbearing potential, a negative pregnancy test must be documented (negative serum pregnancy test performed at the time of screening and negative serum or urine pregnancy test prior to the first dose of study drug)
* The effects of blinatumomab and revumenib on the developing human fetus are unknown. For this reason and because menin inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of blinatumomab and revumenib administration. Males must also agree to refrain from sperm donation during this time period.
* Adequate cardiac function as assessed clinically by history and physical examination with an ejection fraction of >50% by echocardiogram or multigated acquisition (MUGA) scan
* White blood cell (WBC) count below 25,000/uL at the time of enrollment. Participants may receive cytoreduction with dexamethasone and/or cyclophosphamide for cytoreduction
* Estimated glomerular filtration rate (GFR) based on local institutional practice for age appropriate determination by Cockcroft Gault formular for adults, with a GFR>60 ml/min/1.73m2
* For participants having previously received stem cell transplant, at least 60 days must have elapsed, and for prior donor lymphocyte infusion, at least 4 weeks must have elapsed
* For participants having previously received immunotherapy, at least 60 days must have passed
* Weight of at least 40 kg
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Active serious infection not controlled by oral or IV antibiotics
* Active secondary malignancy other than skin cancer (basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Participants with psychiatric illness that would limit compliance with study requirements
* Untreated CNS disease. Participants with controlled CNS disease may be included (as defined by being asymptomatic and having CNS cleared of leukemic involvement)
* Detectable HIV viral load within the previous 6 months. Participants with a known history of HIV must have viral load testing prior to study enrollment.
* Any of the following within 6 months prior to study entry: myocardial infarction, congestive heart failure New York Heart Association Classification Class > II, life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack
* QTc using Friderica's correction (QTcF) >450 msec
* Personal of family history of long QT syndrome
* Cirrhosis with a Child Pugh score of B or C
* Participants with active hepatitis B (defined as Hepatitis B surface antigen with detectable Hepatitis B virus DNA by PCR) or hepatitis C infection (defined as presence of detectable Hepatitis C virus RNA by PCR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05-18 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Elias J Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org